CLINICAL TRIAL: NCT06111690
Title: Feasibility of Prehabilitation Blood-flow Restriction Training in Individuals Awaiting Total Knee Replacement.
Brief Title: Blood Flow Restriction Training in Individuals Awaiting Total Knee Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Gustavo Almeida, Assistant Professor, The University of Texas Health Science Center at San Antonio
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HSC20210590H; 5P30AG044271 (NIH)
Record Dates: First submitted 2023-10-26; First posted 2023-11-01 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Knee Osteoarthritis
Keywords: Blood flow restriction training (BFRT); Preoperative exercise; Muscle function; Physical activity
MeSH Terms: conditions — Osteoarthritis, Knee; Motor Activity | interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Intervention Model Description: This is a single group pre-post design study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Preoperative Exercises (Experimental): Intervention is blood flow restriction training (BFRT)
  Interventions: Procedure: Blood Flow Restriction Training (BFRT)

INTERVENTIONS:
Procedure: Blood Flow Restriction Training (BFRT) — Participants will be performing low-resistance exercise with (BFRT). Intervention will start at least seven days after initial evaluation, so it does not influence measures of real-time physical activity. We will use a log to register exercise completion and to record bilateral knee pain before, during and after each intervention session
  Other Names: BFRT

SUMMARY:
The aim is to demonstrate that preoperative exercises (prehabilitation) using blood-flow restriction training (BFRT) is safe, well tolerated, improves muscle function, decreases functional limitation, and increases physical activity in older adults awaiting total knee replacement (TKR).

DETAILED DESCRIPTION:
Twenty individuals ≥60 years old awaiting TKR due to diagnosis of end-stage knee osteoarthritis who meet the inclusion/exclusion criteria will be invited to participate in a 6 weeks of low-intensity BFRT prehabilitation. We will assess muscle functional (i.e., cross-sectional area and intramuscular fatty content) using computerized tomography, quadriceps muscle strength using an isokinetic dynamometer, a battery of performance-based physical function, self-reported physical function and quality of life, and biomarkers of inflammation using blood serum. Feasibility assessment will be done by looking at safety (i.e., adverse events), compliance, and attrition rate.

ELIGIBILITY:
Inclusion Criteria:

1. Participants are awaiting primary unilateral TKR due to diagnosis of end-stage KOA. Potential individuals must have at least 8 weeks waiting time in between study baseline assessment and surgery. This 8-week timeframe will allow for completion of baseline (T0) and follow-up assessments (T1: immediately after 6-week prehabilitation program);
2. are older than 60 years;
3. speak fluent English to reliably complete the study questionnaires and understand study instructions.

Exclusion Criteria:

1. have a history of cardiovascular disease, uncontrolled hypertension (blood pressure ≥140/90 mmHg), deep-vein thrombosis, varicose veins, or rhabdomyolysis;
2. have absolute contraindications to exercise, as established by the American College of Sports Medicine (uncontrolled arrhythmias, third degree heart block, recent EKG changes, unstable angina, acute myocardial infarction, and acute congestive heart failure);
3. report of 2 or more falls within the past year;
4. cannot walk a distance of 100 feet (30.5 meters) without an assistive device or need of a rest period;
5. have bilateral TKR or undergoing TKR revision or other total joint replacement in the lower extremities; or
6. have severe visual or hearing impairment. In addition to the affects that these impairments have on safety during participation in the intervention, they may also interfere with data collection (questionnaires and telephone checks);
7. have a lower extremity amputation;
8. are unable to comfortably bear weight on the affected knee;
9. have a BMI above 40.
10. history of muscular disease (e.g., muscular dystrophy) or neurological disorder that may affect lower extremity function (e.g., cerebrovascular accident, neuropathy, Parkinson's disease, multiple sclerosis);
11. had additional surgery to the lower extremities within the past 12 months.
12. a Folstein Mini-Mental State Examination score of <24.
13. have acute or terminal illness;
14. are planning to have another TKR (primary on contralateral, or revision on same knee) within 4 months;
15. are planning to relocate to another city within 4 months.
16. Subjects with Sickle cell disease
17. lymphedema or vascular access restrictions
18. Subjects who have any on-going medical emergency
19. An ankle-brachial index outside of the expected range 0.9 and 1.3

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-09-23 (Actual); Primary Completion 2024-10-02 (Actual); Study Completion 2024-12-02 (Actual)

PRIMARY OUTCOMES:
Quadricep Muscle Strength | Baseline, 8 weeks and 16 weeks
  Changes in strength will be measured using an isokinetic dynamometer. Quadriceps femoris maximum voluntary isometric contraction (MVIC) as torque output (Nm) will be measured. Subjects will be seated in the dynamometer's chair with their knee at 60 degrees of flexion.
Thigh muscles composition | Baseline, 8 weeks and 16 weeks
  Change in thigh muscles % fat-free mass and % fat mass will be measured using a DXA scan.
Thigh muscle volume | Baseline, 8 weeks and 16 weeks
  Change in thigh muscles cross-sectional area (volume) will be measured using a DXA scan.

SECONDARY OUTCOMES:
Self-selected Gait Speed | Baseline, 8 weeks and 16 weeks
  Subject will walk a 4-meter walkway at a self-selected pace. Time to complete task will be recorded.
Timed up and go Test | Baseline, 8 weeks and 16 weeks
  Subject will get up from a chair, walk 3 meters, turn around and walk back to and sit on the chair. Time to complete task will be recorded.
30-second chair stand test | Baseline, 8 weeks and 16 weeks
  Subject will perform sit-to-stand from a standard chair for 30 seconds. Number of times of completed sit-to-stand in 30 seconds will be recorded.
Stair climb test | Baseline, 8 weeks and 16 weeks
  Subject will climb up and down a flight of stairs (11 steps). Time to complete task will be recorded.
6-minute Walk Test | Baseline, 8 weeks and 16 weeks
  Subjects will cover as much as they can while walking on a flat, unobstructed path for 6 minutes.
Patient-Reported Physical Outcome | Baseline, 8 weeks and 16 weeks
  Patient-Reported Physical Outcome will be assessed using PROMIS® (Patient-Reported Outcomes Measurement Information System), which is used to evaluate and monitor physical, mental, and social health in persons with several conditions.
Health Related Quality of Life (RAND-36) | Baseline, 8 weeks and 16 weeks
  the RAND-36 Questionnaire is comprised of 36 items that assess eight health concepts: physical functioning, role limitations caused by physical health problems, role limitations caused by emotional problems, social functioning, emotional well-being, energy/fatigue, pain, and general health perceptions.
Real-time Physical Activity | Baseline, 8 weeks and 16 weeks
  An activity monitor will be worn for 7 days and physical activity (i.e., daily number of steps) will be tracked.
Inflammatory Biomarkers | Baseline, 8 weeks and 16 weeks
  Change in 'MILLIPLEX® MAP Human High Sensitivity T Cell Magnetic Bead Panel' to assess a panel of 8 inflammatory biomarkers: Interleukin (IL)-1β, IL-2, IL-5, IL-6, IL-10, IL-12p70, IL-13 and Interferon-γ.

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo Almeida, PhD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- UT Health San Antonio- Dept. of Physical Therapy, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be shared with other researchers at UT Health San Antonio, with the NIH and on ClinicalTrials.gov
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will become available after summary result publication on ClinicalTrials.gov and when published in a peer review journal